CLINICAL TRIAL: NCT03360058
Title: Obesity and Type 2 Diabetes - Raising the Issue of Weight Management in Primary Care (Small Talk Big Difference)
Brief Title: Obesity and Type 2 Diabetes - Raising the Issue of Weight Management in Primary Care
Acronym: STBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GN17DI319
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Weight Management; Diabetes Mellitus, Type 2
Keywords: motivational techniques; primary care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Primary care practices are either assigned to immediate or delayed access to the online training and print pieces with the delayed group acting as our controls for number of referral to weight management services per practice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate access to STBD training (Experimental): Immediate access to training materials and print pieces to support implementation
  Interventions: Behavioral: Small Talk Big Difference Immediate access training
- Delayed access to STBD training (Placebo Comparator): Delayed access to training materials and print pieces
  Interventions: Behavioral: Small Talk Big Difference delayed access training

INTERVENTIONS:
Behavioral: Small Talk Big Difference Immediate access training — Immediate access to 1 hour online training and supporting print materials for implementation in primary care practice
  Arms: Immediate access to STBD training
Behavioral: Small Talk Big Difference delayed access training — Delayed access (by 4 months) to 1 hour online training and supporting print materials for implementation in primary care practice
  Arms: Delayed access to STBD training

SUMMARY:
To ensure that patients who are overweight or obese and have type 2 diabetes are identified, receive personalised diabetes care, have the issue of weight raised and explained in a non-judgemental manner by staff in primary care, and are referred on to weight management services as appropriate ensuring equity of access across NHS Greater Glasgow and Clyde.

Specific aims of the whole project:

1. To improve GP/ primary care staff knowledge of the evidence base for the management of diabetes when there is co-existing obesity and local care pathways
2. To increase GP/ primary care staff knowledge of and confidence in their role in raising the issue of weight management,
3. To improve primary care referral rates of appropriate patients who are overweight or obese and have type 2 diabetes, and are "ready to change" to NHS funded weight management services
4. To improve patient uptake of and attendance at NHS funded weight management services NB This is a service evaluation of a training programme being delivered by NHS Greater Glasgow and Clyde Health Improvement. Full ethical approvals are being sought due to the randomised design and so that results can be generalised and published.

DETAILED DESCRIPTION:
The Glasgow and Clyde weight management service (GCWMS) delivers a specialist multi-disciplinary, multi-component weight management programme throughout the Glasgow and Clyde area. In a recent evaluation of the service, the authors highlighted that 27% of the patients who are referred to the programme do not opt into the service. This describes patients who are referred via their GP practice and do not contact the service to opt into an initial assessment.

Similarly, Brook et al described initial uptake and engagement of a small weight management programme of 502 patients. In addition to completing an extensive questionnaire, patients were requested to call to make an appointment with the service personally. Of those referred to the programme, 46% did not opt in.

Engaging patients in a weight management programme is especially difficult, even when the intervention is provided via the primary care route. For example, The Counterweight Project, a weight management programme delivered via the GP surgery, has been taken up by a number of surgeries in Scotland, however after 2 years, one fifth of enlisted practices failed to enrol patients onto the programme.

Even when GP's do address matters of weight related behaviour, there is often disagreement from the patient that the topic has been raised. In a sample of 456 patients, 39% of patients disagreed with GP reporting about the content of the discussion during consultations regarding weight, diet and physical activity. In particular, GP's reported more occasions of discussing weight than patients in 12.5% of consultations. Patients' likeliness to engage in a weight management programme is also influenced by practice endorsement and opinion of the GP of the intervention available in addition to other factors: clear understanding of the programme, clear understanding of the programme goals, structured pro-active follow-up and perception of positive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* GP practices in NHS Greater Glasgow and Clyde which:
* Have a contract for local enhanced services for long term conditions (Diabetes)
* Have a unique clinical database (i.e. not shared with another practice)

Exclusion Criteria:

* "17c" practices (those with a separate contract for long term conditions)
* Those practices with a database shared with another practice (8 practices in area)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-07 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Measure the effectiveness of an online training programme, practice implementation toolkit and face to face training for primary care staff | 12 months
  which will be measured as number of patient referrals and patient attendance at NHS funded weight management services

SECONDARY OUTCOMES:
Implementation/ Normalization | 12 months
  NOMAD questionnaire will be used to ascertain how STBD impacts on primary care clinicians work
Percentage of diabetes reviews with recorded weight management discussion in LES template | 12 months
  percentage of diabetes review in primary care
Training uptake | 12 months
  Training uptake - online, face to face and experiential
  * By practice
  * By GP and practice Nurse By diabetes lead

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Logue, MBChB PhD, Principal Investigator — Glasgow University and NHS GGC
Locations (1):
- Glasgow Cardiovascular Research Centre, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brooksbank K, O'Donnell J, Corbett V, Shield S, Ainsworth R, Shearer R, Montgomery S, Gallagher A, Duncan H, Hamilton L, Laszlo V, Noone R, Baxendale A, Blane D, Logue J. Discussing Weight Management With Type 2 Diabetes Patients in Primary Care Using the Small Talk Big Difference Intervention: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Feb 15;8(2):e12162. doi: 10.2196/12162. PMID 30767902